CLINICAL TRIAL: NCT04037241
Title: A Randomized Open-Label Phase 2b Study of Hepatic Infusions of Anti-CEA CAR-T Cells Alternating With Systemic Chemotherapy Versus Chemotherapy Alone In Patients With Liver Metastases Due To CEA-Expressing Pancreatic Adenocarcinoma
Brief Title: Study of Anti-CEA CAR-T + Chemotherapy VS Chemotherapy Alone in Patients With CEA+Pancreatic Cancer & Liver Metastases
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STI-CEA-201
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Malignant Tumor of Pancreas Metastatic to Liver
MeSH Terms: interventions — Gemcitabine; Albumin-Bound Paclitaxel; irinotecan sucrosofate; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 2nd Line: Anti-CEA CAR-T Cells + gemcitabine/nab paclitaxel (Experimental): Patients in the "anti-CEA CAR-T Cells plus gemcitabine/nab paclitaxel arm" will have achieved at least stable disease during the Bridging Therapy Period with gemcitabine/nab paclitaxel, and will receive the CAR-T cells in Cycles 1 and 3 and the gemcitabine/nab paclitaxel regimen they received during the Bridging Therapy Period in Cycle 2 and Cycles ≥ 4 of the Treatment Period. Treatment will continue until the development of disease progression.
  Interventions: Biological: Anti-CEA CAR-T cells; Drug: gemcitabine/nab paclitaxel
- 2nd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA (Experimental): Patients in the "anti-CEA CAR-T Cells plus and nanolipsomal irinotecan (NLIR) + Fluorouracil/folinic acid (FU/FA)" will have achieved at least stable disease during the Bridging Therapy Period with NLIR + FU/FA, and will receive the CAR-T cells in Cycles 1 and 3 and the NLIR/FU/FA regimen they received during the Bridging Therapy Period in Cycle 2 and Cycles ≥ 4 of the Treatment Period. Treatment will continue until the development of disease progression.
  Interventions: Biological: Anti-CEA CAR-T cells; Drug: NLIR+FU/FA
- 2nd Line: Gemcitabine /nab paclitaxel Alone (Active Comparator): Patients in the chemotherapy alone treatment arm who achieved at least stable disease during the Bridging Therapy Period while receiving gemcitabine plus nab paclitaxel will continue treatment with the chemotherapy regimen they received during the Treatment Period. This regimen will be administered in 28-day cycles until the development of disease progression.
  Interventions: Drug: gemcitabine/nab paclitaxel
- 2nd Line: NLIR + FU/FA Alone (Active Comparator): Patients in the chemotherapy alone treatment arm who achieved at least stable disease during the Bridging Therapy Period while receiving nanoliposomal irinotecan (NLIR) + Fluorouracil/folinic acid (FU/FA) will continue treatment with the chemotherapy regimen they received during the Treatment Period. This regimen will be administered in 28-day cycles until the development of disease progression.
  Interventions: Drug: NLIR+FU/FA
- 3rd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA (Experimental): Patients randomized to the anti-CEA CAR-T Cells plus chemotherapy treatment arm who developed disease progression during the Bridging Therapy Period will receive the CAR-T cells in Cycles 1 and 3. Nanoliposomal irinotecan plus fluorouracil/leucovorin chemotherapy will be administered in Cycle 2 and Cycles ≥ 4 of the Treatment Period to patients who progressed on nab paclitaxel plus gemcitabine during the Bridging Therapy Period. Treatment will continue until the development of disease progression.
  Interventions: Biological: Anti-CEA CAR-T cells; Drug: NLIR+FU/FA
- 3rd Line: Anti-CEA CAR-T Cells Plus Capecitabine (Experimental): Patients randomized to the anti-CEA CAR-T Cells plus chemotherapy treatment arm who developed disease progression during the Bridging Therapy Period will receive the CAR-T cells in Cycles 1 and 3. Capecitabine chemotherapy will be administered in Cycle 2 and Cycles ≥ 4 of the Treatment Period to patients who progressed on nanoliposomal irinotecan fluorouracil/leucovorin during the Bridging Therapy Period. Treatment will continue until the development of disease progression.
  Interventions: Biological: Anti-CEA CAR-T cells; Drug: Capecitabine
- 3rd Line: NLIR+FU/FA Alone (Active Comparator): Patients randomized to the chemotherapy alone treatment arm who developed disease progression during the Bridging Therapy Period while receiving nab paclitaxel plus gemcitabine will be treated with nanoliposomal irinotecan plus fluorouracil/leucovorin during the Treatment Period.
  Interventions: Drug: NLIR+FU/FA
- 3rd Line: Capecitabine Alone (Active Comparator): Patients that developed disease progression during the Bridging Therapy Period while receiving nanoliposomal irinotecan plus 5-FU/leucovorin will be treated with capecitabine during the Treatment Period.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Biological: Anti-CEA CAR-T cells — Doses will be delivered by hepatic arterial infusions using a pressure enabled drug delivery (PEDD) device
  Other Names: SureFire Precision Infusion System; K171355; TriSalus PEDD
  Arms: 2nd Line: Anti-CEA CAR-T Cells + gemcitabine/nab paclitaxel; 2nd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA; 3rd Line: Anti-CEA CAR-T Cells Plus Capecitabine; 3rd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA
Drug: gemcitabine/nab paclitaxel — systemic chemotherapy regimen
  Other Names: Gemzar; Abraxane
  Arms: 2nd Line: Anti-CEA CAR-T Cells + gemcitabine/nab paclitaxel; 2nd Line: Gemcitabine /nab paclitaxel Alone
Drug: NLIR+FU/FA — systemic chemotherapy regimen
  Other Names: Onivyde; Adrucil; Leucovorin
  Arms: 2nd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA; 2nd Line: NLIR + FU/FA Alone; 3rd Line: Anti-CEA CAR-T Cells Plus NLIR+FU/FA; 3rd Line: NLIR+FU/FA Alone
Drug: Capecitabine — systemic chemotherapy regimen
  Other Names: Xeloda
  Arms: 3rd Line: Anti-CEA CAR-T Cells Plus Capecitabine; 3rd Line: Capecitabine Alone

SUMMARY:
This study is a randomized open-label phase 2b study of the efficacy and safety of regional infusion therapy with Anti-CEA CAR-T cells using the hepatic immunotherapy for metastases (HITM) method and the Trisalus pressure enabling drug delivery (PEDD) device alternating with systemic chemotherapy versus chemotherapy alone in patients with CEA-expressing pancreatic adenocarcinoma with liver metastases.

DETAILED DESCRIPTION:
The study consists of 5 periods: Screening/Leukapheresis Period, Bridging Therapy Period, Randomization Period, Treatment Period, and Observation Period (which will be the long-term follow-up period to monitor for overall survival and long-term safety).

Patients in this trial with CEA-expressing pancreatic adenocarcinoma with liver metastases must have developed disease progression after first-line treatment with FOLFIRINOX (irinotecan, 5-fluorouracil, leucovorin, and oxaliplatin) or gemcitabine-based chemotherapy. Patients will be randomized to either the "anti-CEA CAR-T Cells + systemic chemotherapy treatment arms", or the "chemotherapy alone treatment arms."

If the patients achieve at least stable disease during the Bridging Therapy Period, they will be in the Second-Line Group of Treatment Arms. Patients who develop disease progression during the Bridging Period will be in the Third-Line Group of Treatment Arms.

Patients in the Second-Line or Third-Line treatment arms who are randomized to the treatment arms of "Anti-CEA CAR-T cells plus systemic chemotherapy" will receive hepatic infusions of Anti-CEA CAR-T cells in Cycles 1 and 3 (ie, each 42-day cycle is 3 weekly doses of Anti-CEA CAR-T cells administered as hepatic arterial infusions using a PEDD device with low dose systemic IL-2 support), alternating with the systemic chemotherapy regimen they received during the Bridging Therapy Period in Cycle 2 and Cycles >= 4. Systemic chemotherapy will be administered in 28-day cycles until the development of disease progression.

Patients in the Second-Line or Third-Line treatment arms who are randomized to the treatment arms "chemotherapy alone" arms will continue to receive the same systemic chemotherapy that they received during the Bridging Therapy Period. Systemic chemotherapy will be administered in 28-day or 21-day cycles (depending on the type of systemic chemotherapy regimen the patient will receive) until the development of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented CEA-expressing pancreatic adenocarcinoma with unresectable liver metastases. Documentation of CEA-expressing adenocarcinoma may be demonstrated by an elevated serum CEA level (≥ 10 ng/mL) or by the detection of CEA on the cell surface of adenocarcino3.
* Documentation of disease progression of pancreatic adenocarcinoma following the initiation of first-line treatment with FOLFIRINOX or gemcitabine-based therapy.ma cells by immunohistochemistry (IHC).
* The primary pancreatic tumor may be intact and limited lung metastases (≤ 3 lesions, none > 1 cm in longest diameter) and lymphoid metastases (≤ 3 lesions, none > 1 cm in longest diameter) are permitted.
* There must be at least one measurable metastatic liver lesion ( ≥ 10 mm in longest diameter).
* ECOG performance status of 0 or 1.
* Be willing and able to comply with the study schedule and all other protocol requirements.
* Females of childbearing potential must have 2 negative pregnancy tests prior to the start of study treatment, and must agree to pregnancy tests during the study; sexually active female and male patients must be willing to use an effective birth control to avoid pregnancy.

Exclusion Criteria:

* Received anti-cancer chemotherapy or investigational systemic anti-cancer treatments other than first line FOLFIRINOX or gemcitabine-based chemotherapy for advanced pancreatic adenocarcinoma.
* Received FOLFIRINOX or gemcitabine-based therapy within 14 days before receiving the first dose of study treatment.
* Have any unresolved toxicity > Grade 1 from previous anticancer therapy, except for stable chronic toxicities (≤ Grade 2) that are not expected to resolve.
* Have a history of histologically confirmed metastases outside the liver, lungs, or lymph nodes.
* More than 50% replacement of one or both hepatic lobes with tumor.
* Tumor causing biliary obstruction not amenable to stenting.
* Received prior anti-CEA agents, CAR-T, CAR-T cell line, CAR-NK, CAR-pNK, or CAR-NK cell line therapies.
* Have any clinically significant low baseline lab results for hemoglobin, platelet counts, or neutrophil counts at screening.
* Has any untreated or ongoing intra-abdominal infection or bowel obstruction.
* Has any clinically significant elevated baseline lab results for serum creatinine, aspartate aminotransferase (AST), and total bilirubin (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome), and alkaline phosphatase at screening.
* Known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C.
* Female patients who are pregnant or breastfeeding.
* Has active bacterial, viral or fungal infections.
* Has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
* Has any condition, including the presence of laboratory abnormalities that places the patient at an unacceptable risk if the patient was to participate in the study.
* Are receiving medications that are strong inducers CYP3A4 or CYP2C8 within 2 weeks of initiating treatment in the Bridging Therapy Period (rifampicin, carbamazepine, phenytoin, efavirenz, nevirapine, rifabutin, rifapentine, St. John's wort).
* Are receiving medications that inhibit CYP3A4 or CYP2C8 within 1 week of initiating treatment in the Bridging Therapy Period (ketoconazole and other imidazole antifungals, erythromycin, clarithromycin, itraconazole, voriconazole, fluoxetine, gemfibrozil, cimetidine, lopinavir, nefazodone, telaprevir, ritonavir, saquinavir, indinavir, or nelfinavir).
* Are receiving medications that inhibit UGT1A1 within 1 week of initiating nanoliposomal irinotecan therapy (atazanavir, gemfibrozil, indinavir).
* Left ventricular ejection fraction (LVEF) < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy by overall survival | 6 - 12 months
  As a measure of activity, Overall Survival (OS) will be assessed. The events for the assessment of OS are death events. Time to event endpoints will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where applicable.

SECONDARY OUTCOMES:
Assess safety by monitoring adverse events | 6 - 12 months
  As a measure of safety, the types, frequencies, and severities of adverse events and their relationship to study drug will be summarized.
Assess efficacy by within-liver progression free survival (PFS) | 6 - 12 months
  As a measure of activity, within-liver PFS will be assessed. The events for the assessment of within-liver PFS will be measured from the date of randomization to the date of disease progression within the liver or death, whichever comes first. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
Assess efficacy by progression free survival (PFS) | 6 - 12 months
  As a measure of activity, PFS will be assessed. The events for the assessment of PFS will be measured from the date of randomization to the date of disease progression or death, whichever comes first. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
Assess efficacy by within-liver time to progression (TTP) | 6 - 12 months
  As a measure of activity, within-liver TTP will be assessed. The events for the assessment of within-liver TTP will be measured from the date of randomization to the date of disease progression within the liver. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
Assess efficacy by time to progression (TTP) | 6 - 12 months
  As a measure of activity, TTP will be assessed. The events for the assessment of TTP will be measured from the date of randomization to the date of disease progression. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where appropriate.
Assess efficacy by within-liver radiographic response rate using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | 6 - 12 months
  As a measure of activity, overall response rate within-liver will be assessed using radiographic scans using RECIST v 1.1 criteria. Response will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Assess efficacy by overall whole-body radiographic response rate using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | 6 - 12 months
  As a measure of activity, overall response rate for overall whole-body will be assessed using radiographic scans using RECIST v 1.1 criteria. Response will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Assess efficacy by duration of response within-liver in accordance with RECIST v 1.1 criteria | 6 - 12 months
  As a measure of activity, duration of response within-liver will be measured using radiologic scans and assessed according to RECIST v1.1 criteria. This will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Assess efficacy by duration of response of overall whole-body in accordance with RECIST v 1.1 criteria | 6 - 12 months
  As a measure of activity, duration of response of overall whole-body will be measured using radiologic scans and assessed according to RECIST v1.1 criteria. This will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Assess efficacy by serologic response rates by CEA levels | 6 - 12 months
  As a measure of activity, overall response rate will be assessed by serologic CEA levels. Response rate will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Assess efficacy by serologic response rates by CA 19-9 levels | 6 - 12 months
  As a measure of activity, overall response rate will be assessed by serologic CA 19-9 levels. Response rate will be assessed for each patient over a 6- to 12-month timeframe during the Treatment and Observation Periods of the protocol.
Evaluation of Quality-of-Life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | 6 - 12 months
  As a measure of quality-of-life, the EORTC QLQ-C30 instrument will be administered at months 2, 4, 6 of the Treatment Period and at the end of study.
Evaluation of Quality-of-Life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Pancreatic Cancer Module (EORTC QLQ-PAN26) | 6 - 12 months
  As a measure of quality-of-life specific for patients with pancreatic cancer, the EORTC QLQ-PAN26 instrument will be administered at months 2, 4, 6 of the Treatment Period and at the end of study.
Evaluation of Quality-of-Life using the 5-level EQ-5D version (EQ-5D-5L) questionnaire | 6 - 12 months
  As a measure of quality-of-life, the EQ-5D-5L questionnaire will be administered at months 2, 4, 6 of the Treatment Period and at the end of study.

OTHER OUTCOMES:
Assess if serum cytokine levels correlate with response and/or toxicity to hepatic arterial infusions | 6 - 12 months
  As an exploratory analysis, serum cytokine levels (pg/mL) will be measured over time by a standard laboratory test using Enzyme-linked immunosorbent assay (ELISA) to determine if increases in cytokines predict response and/or toxicity to liver arterial infusions.
Assess if neutrophil: lymphocyte ratio (NLR) correlate with response from hepatic arterial infusions | 6 - 12 months
  As an exploratory analysis, NLR will be calculated to determine if there is a correlation with response and/or toxicity.
Assess the persistence of CAR-T cells in liver tumor biopsies over time. | 6 - 12 months
  As an exploratory analysis, the engraftment of CAR-T cells in planned liver tumor biopsies will be analyzed to assess persistence of CAR-T cells during the Treatment and Observation Periods of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yan, MD MS, Study Director — Sorrento Therapeutics